CLINICAL TRIAL: NCT03531788
Title: Use of Dynamic Arm Support Devices for Upper Limb Function in Non-Ambulatory Men With Duchenne Muscular Dystrophy (DMD)
Brief Title: Use of Dynamic Arm Supports to Promote Activities of Daily Living in Individuals With DMD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID inhibited additional home visits for device installation and testing
Sponsor: Roxanna Marie Bendixen (Other)
Responsible Party: Sponsor-Investigator, Roxanna Marie Bendixen, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO18010005
Record Dates: First submitted 2018-04-02; First posted 2018-05-22 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: dynamic arm support; mobile arm support; rehabilitation; occupational therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to trial a dynamic arm support (Armon Ayura (Kinova) or JAECO WREX)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Armon Ayura (Kinova) (Experimental): Participants will trial the Armon Ayura dynamic arm support.
  Interventions: Device: Armon Ayura (Kinova)
- JAECO WREX (Experimental): Participants will trial the JAECO Wilmington Robotic EXoskeleton (WREX) dynamic arm support.
  Interventions: Device: JAECO Wrex

INTERVENTIONS:
Device: Armon Ayura (Kinova) — Actively assisted mechanical arm support (electric powered to balance arm)
  Other Names: Kinova
  Arms: Armon Ayura (Kinova)
Device: JAECO Wrex — Passive mechanical arm support (elastic bands to balance arm)
  Arms: JAECO WREX

SUMMARY:
This study is a longitudinal, randomized control trial evaluating the use of two commercially available dynamic arm support devices (1) Armon Ayura-Kinova and 2) JAECO WREX) to promote participation in activities of daily living (ADLs) in non-ambulatory individuals with Duchenne muscular dystrophy (DMD) with upper extremity weakness.

DETAILED DESCRIPTION:
This study is a longitudinal, randomized control trial evaluating the use of two commercially available dynamic arm support devices (1) Armon Ayura-Kinova and 2) JAECO WREX) to promote participation in activities of daily living (ADLs) in non-ambulatory individuals with Duchenne muscular dystrophy (DMD) with upper extremity weakness. Up to 30 individuals will be enrolled to participate in this research study, which includes a two-week baseline data collection period, a four-week device trial and a two-week post device data collection period. Participants will be randomly assigned to trial one of the dynamic arm support devices during the four week in-home trial. The ActiGraph GT9x (name of device), a wrist worn activity monitoring device, will be worn during the baseline period, the device trial and the post device data collection period to capture upper extremity (UE) movement patterns. UE performance will be further quantified with use of a physical motor assessment, the Performance of Upper Limb (PUL) assessment and patient reported outcomes. Data gleaned will provide important knowledge and objective results regarding the potential benefit of dynamic arm supports in individuals with DMD with limited functional use of their upper extremities.

ELIGIBILITY:
Inclusion Criteria:

1. 14 years of age or older
2. Self-report diagnosis of Duchenne muscular dystrophy (DMD)
3. Use a wheelchair for mobility
4. Score 3-5 on the Brooke Upper Extremity (UE) Scale
5. Self-report of needs assistance/unable to achieve independently on at least 10 items on the Upper Limb Activities of Daily Living (UL ADL) self-report questionnaire
6. Able to follow instructions
7. Informed consent provided by self (18 and over) or by parent or legal guardian (if under the age of 18)

Exclusion Criteria:

1. Does not have minimum level of UE function to operate the assigned dynamic arm support (Score of 6 on the Brooke UE scale or any other impairment limiting use)
2. The assigned dynamic arm support is unable to be mounted to wheelchair (mounts will vary based on manufacturer/model of wheelchair)

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxanna M Bendixen, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Armon Ayura (Kinova) | JAECO WREX
Started | 12 | 6
Completed | 11 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armon Ayura (Kinova) | JAECO WREX | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.10 (2.32) | 18.22 (4.20) | 18.16 (3.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18
Actigraphy (wrist worn activity monitor) [Mean (Standard Deviation); unit: activity counts] — Baseline data were collected using wrist worn Actigraph GT9x during baseline assessment of upper extremity function without the dynamic arm support device. Data were collected over a 2-week time period and means and standard deviation activity counts were used. Actigraph GT9x provides activity counts which measure movement in all directions. Population: Data were collected using wrist worn Actigraph GT9x during baseline assessment of upper extremity function without the dynamic arm support device. Data were collected over a 2-week time period and means and standard deviation activity counts were used. Actigraph GT9x provides activity counts which measure movement in all directions. The Actigraph was not worn during baseline testing for some participants, resulting in missing activity count data. Higher activity counts represents more movement.
  activity counts
    number analyzed (Participants) | 7 | 3 | 10
    (all) | 534.02 (321.35) | 235.80 (150.51) | 444.55 (307.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Activity Counts (Movement) Through Actigraphy
Description: Measured through the ActiGraph GT9X wrist worn activity monitoring device: The multi-axis activity monitor measures activity counts that represent movement of the upper extremity. We calculated the average activity counts during testing items with the arm device and testing items without the arm device. We then calculated change scores (average activity counts without the device minus average activity counts with the device). Higher activity counts indicate more effort and more movement during item testing without the device compared to using the device.
Time Frame: Collection of activity counts through the ActiGraph GT9x occurred during testing phase with and without the upper extremity arm device.
Population: All participants who had completed the testing period while wearing the Actigraph GT9x are reported. All participants were tested, but data are missing due to technology failure or not wearing the ActiGraph during testing. Participants who were not wearing the ActiGraph during testing are not reported. Comparisons between groups (Kinova and WREX) were not analyzed due to small sample sizes in both groups.
Measure: Mean (Standard Deviation); unit: Activity Counts
Arm/Group | Armon Ayura (Kinova) | JAECO WREX
Number analyzed (Participants) | 7 | 3
Activity Counts | 270.61 (375.50) | 26.75 (123.04)
Statistical Analysis 1: Comparison: Armon Ayura (Kinova) vs JAECO WREX; Activity counts from the ActiGraph GT9x activity monitor provide data per participant during testing of upper extremity activities/tasks and were collected while wearing the device (Kinova and WREX) and without the device (Kinova and WREX). For each upper extremity task, we summed all activity count data for all tasks completed. We then computed means and standard deviations. Data presented are within group data change and not between group data comparisons; Test type: Other; Due to the small sample size, we utilized change in activity count data when comparing two upper limb testing sessions: one without the use of an arm support device (Kinova or WREX) and one while using the arm support device. For each upper extremity task, we summed all activity count data for all tasks completed. We then computed means and standard deviations. Data presented are within group data change and not between group data comparisons

2. Primary Outcome: Change in Upper Extremity Position Through Actigraphy
Description: Measured through the ActiGraph GT9X wrist worn activity monitoring device: The multi-axis activity monitor (gyroscope within the monitor) measures activity counts (movement) per second in the x, y, and z planes. Change in average activity counts (movement) in x, y, and z planes during the 4-week trial period compared to the 2-week baseline period are reported (higher activity counts means more movement during trial). X plane is horizontal movement, y plane is vertical movement, and z plane extends outward from the body.
Time Frame: Collection of activity counts through the ActiGraph GT9x occurs from baseline through the end of the 4-week device trial.
Population: All participants who completed the testing period while wearing the Actigraph are reported. Comparisons between groups (Kinova and WREX) were not analyzed due to small sample sizes in both groups.
Measure: Mean (Standard Deviation); unit: Activity Counts
Arm/Group | Armon Ayura (Kinova) | JAECO WREX
Number analyzed (Participants) | 10 | 4
Activity Counts
  Average x axis change score | 19838.12 (41880.09) | 44697.80 (89132.49)
  Average y axis change score | 69125.26 (102942.92) | 1279.76 (141962.15)
  Average z axis change score | 59784.84 (91039.70) | 17297.11 (130688.29)
Statistical Analysis 1: Comparison: Armon Ayura (Kinova) vs JAECO WREX; Activity counts from the ActiGraph GT9x activity monitor were collected during baseline (without a device) and throughout the 4 week device trial (with the device). For each time period, activity count data were averaged across the day. We then compared the baseline time period to the device trial period to understand the difference in movement and upper extremity positioning during the device trial. Data presented are within group change scores and not between group data comparisons; Test type: Other; Counts from each axis (x, y, z) were measured across baseline and during the 4-week trial to explore arm movement and positioning during the use of an upper extremity arm device. Counts (within each participant) were summed. A change score from trial minus baseline was calculated for each axis. We provide an average change score and standard deviation across participants with Kinova and participants with WREX

3. Secondary Outcome: Goal Attainment Scale (GAS)
Description: The GAS is a personal interview which allows the individual to determine important and personally meaningful goals. Each participant chose three individualized goals to work on and assess at the end of the study. Goal scaling is standardized in order to calculate the extent to which a patient's goals are met.The GAS uses a 5-point rating scale to determine if the goal was not met (-2) up to a greater than expected meeting of the personal goal (+2). A score of 0 indicates the goal was met as anticipated. We report the average change in the score of each goal when the participant uses the trial device. Here we use change scores which range from 0 (performed the same with and without the device) to 4 (participant performed at a greater than expected level with the device).
Time Frame: The GAS is completed and scored at baseline and at the end of the 4 week trial with and without the device.
Population: Participants were included in this analysis if they completed the Goal Attainment Scale (GAS) with and without the use of the arm device (Kinova or WREX). Sample sizes were too small to use statistical analyses for comparisons between groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Armon Ayura (Kinova) | JAECO WREX
Number analyzed (Participants) | 11 | 4
score on a scale
  Goal 1 | 3.09 (0.83) | 3.5 (1.0)
  Goal 2 | 2.72 (1.9) | 2.75 (1.9)
  Goal 3 | 3.18 (0.87) | 3.5 (0.58)
Statistical Analysis 1: Comparison: Armon Ayura (Kinova) vs JAECO WREX; Three goals were identified for each participant and scored without using an arm support device to serve as a baseline measure of abilities. These scores were compared to the scores achieved on the same goals using the arm support device; Test type: Other; We compared the change in GAS scores when using an arm support device on three goal areas identified as important for each participant. For each goal, we measured abilities at baseline and with the device (Kinova and WREX). We calculated the change in score for each goal and averaged these change scores across all participants. While our groups are too small to complete statistical tests to estimate the significance of the differences participants noted in activity and independence while using both arm supports, our results quantify the amount of increased success participants noted with the use of the arm support device

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected for up to 10 weeks.
Description: Participants were monitored throughout baseline data collection, the 4 week in-home device trial, and 2 weeks following the removal of the arm device. We maintained contact with participants throughout the study and recorded any adverse or serious adverse event.
Arm/Group | Armon Ayura (Kinova) | JAECO WREX
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 0/6

LIMITATIONS AND CAVEATS:
Coronavirus disease 2019 (COVID) occurred during recruitment and testing, which required us to terminate the trial early before achieving full recruitment. Technical problems with the accelerometer (Actigraph GT9x) led to missing data. At times testing occurred when the participant was not wearing the accelerometer, also leading to missing data. Sample sizes were therefore too small to compute p values or provide any comparative data (between devices). Therefore, change scores were recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03531788/Prot_SAP_001.pdf